CLINICAL TRIAL: NCT05745506
Title: Effect of Sleep Disorder on the Development of Lung Tumors, a Perspective, Single-centered Study
Brief Title: Effect of Sleep Disorder on the Development of Lung Tumors
Status: Not yet recruiting | Type: Observational
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IIT-2022-0160
Record Dates: First submitted 2023-02-16; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Sleep Disorder, Lung Tumor
MeSH Terms: conditions — Sleep Wake Disorders; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — lung tumor tissue from sublobectomy

GROUPS / COHORTS (2):
- CRD: patients whose PSQI score>5
- non-CRD: patients whose PSQI score ≦ 5

INTERVENTIONS:
Other:  — Not applicable, there is no intervention description in this study.

SUMMARY:
The goal of this observational study is to observe the lung tumor development in lung tumor patients with long-term sleep disorder. The main questions it aims to answer are:

* will long-term sleep disorder promote the malignancy of lung tumor
* if so, how exactly will the microenvironment of lung tumor change Participants will receive PSQI scale and MRI functional brain imaging before surgery, blood and tumor tissue will be collected during the surgery.

Researchers will set non-sleep disorder group as control group to see if lung tumor microenvironment change when long-term sleep disorder exists in lung tumor patiens.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* elective sublobectomy for primary lung tumor
* ASA grade I-II
* Informed consent of the patient or family

Exclusion Criteria:

* Combination of serious heart, liver, kidney, central nervous system, blood system, immune system diseases or serious mental illness
* Combination of other cancers
* untreated active lung infection
* patients with preoperative neoadjuvant radiotherapy

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants are 18-75 years old man or women diagnosed with primary lung tumor.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
tumor microenvironment in sleep-disordered lung cancer patients | 3 months after surgery
  we use single cell sequencing to analyze microenvironment alterations of tumor tissues in enrolled patients.

SECONDARY OUTCOMES:
peripheral blood levels of neurotransmitters in sleep-disordered lung cancer patients | 3 months after surgery
  peripheral blood levels of epinephrine, noradrenaline, 5-HT in sleep-disordered lung cancer patients
Functional brain imaging in sleep-disordered lung cancer patients | 3 months after surgery
  Functional brain imaging

CONTACTS AND LOCATIONS:
Overall Officials: Weifeng Yu, Study Director — Department of Anesthesiology, Renji Hospital, Shanghai Jiaotong University School of Medicine

IPD SHARING:
Plan to Share IPD: Undecided